CLINICAL TRIAL: NCT05240937
Title: The Effect of Mindfulness-Based Self-Compassion Program on Ontological Well-Being Levels of Breast Cancer Patients
Brief Title: The Effect of Self-compassion on Breast Cancer
Acronym: cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Behice Belkıs ÇALIŞKAN, Researcher, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/32
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Self Compassion
Keywords: Mindfulness; Self Compassion; ontological well-being
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based self-compassion will be applied (Experimental): The group in which mindfulness-based self-compassion program will be implemented.
  Interventions: Behavioral: mindfulness-based self-compassion will be applied
- Control Group (No Intervention): The group in which mindfulness-based self-compassion program will not be implemented

INTERVENTIONS:
Behavioral: mindfulness-based self-compassion will be applied — A mindfulness-based self-compassion program will be applied to this group of patients who have had breast cancer and have fully completed their treatment.
  Arms: mindfulness-based self-compassion will be applied

SUMMARY:
Most women don't want to hear the word cancer, so they feel anxious and stressed. However, "cancer" can be the beginning of learning how to fight and being hopeful. Ontological well-being is a concept that includes the life project of the individual and the meaning of life. the life of the individual; It is a project that includes the past tense, present tense and future tense components. Mindfulness-based practices are an application that examines the psychological and physiological aspects of stress and includes the concept of self-compassion. Self-compassion requires a balanced approach to one's negative emotions. When studies with breast cancer patients are examined, it is emphasized that self-compassion has an effect on concepts such as quality of life, anxiety, depression, and body image. This research was planned to determine the effectiveness of the awareness-based self-compassion program applied to patients with breast cancer on the ontological well-being of individuals.

DETAILED DESCRIPTION:
Research Design Research; In order to determine the effect of the mindfulness-based self-compassion program to be applied to patients with breast cancer on the oncological well-being of individuals, it was planned as a randomized controlled study with a pretest-posttest control group.

Research Hypotheses H1: The scores of breast cancer patients participating in the mindfulness-based self-compassion program will increase in the ontological well-being scale.

Place and Time of Research The research will be carried out at Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty Hospital between February 2022 and September 2022.

Population and Sample of the Research The population of the research will consist of individuals who were diagnosed with breast cancer, completed their treatment and are in the follow-up phase in Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty Hospital.

The sample of the study will consist of at least 70 individuals determined by power analysis.

Randomization: A pre-test will be done by pre-interviewing the patients, and patients with a maximum score of 25 on the Beck Depression Scale and patients who meet the inclusion criteria will be included in the study. Computer-assisted randomization will be performed by an independent statistician according to the list of patients who meet the inclusion criteria.

In this study, the scales will be applied as Pre-Post-Test. It does not pose any problem that will endanger the physical and mental health of the participants.

* Individual Characteristics Form
* Ontological Well-Being Scale (OWBS)
* Beck Depression Scale (BDI)

An 8-week Awareness-Based Self-Compassion Program will be applied to the experimental group determined according to the randomization results. After the application, the experimental and control groups will be given a post-test and followed up 3 months later. A mindfulness-based self-compassion program will be applied to the control group after the application is made to the experimental group and after the study is completely finished.

Expected Benefit and Widespread Effect By implementing the Awareness-Based Self-Compassion Program, by affecting the ontological well-being of patients who have overcome breast cancer and are in the control phase, discovering the meaning and purpose of life, to look at life with hope, keep motivation high for the present It is aimed to increase the sense of satisfaction related to the quality of life of the individual arising from his own self.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with breast cancer
* Being in the control process that has completed the treatment process
* Having a score of 0-25 on the Beck Depression Scale
* Not having a psychiatric diagnosis and no treatment
* be between the ages of 30-55
* Being a literate writer
* Being able to use the internet and social media easily

Exclusion Criteria:

* be in treatment
* Having a score above 25 on the Beck Depression Scale
* Having a psychiatric diagnosis and history
* to be illiterate

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since the incidence of breast cancer in women is very high, the study will be conducted for women.
Enrollment: 70 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Ontological Well Being Scale | 8 Months
  Ontological Well-Being (OWB) is a concept introduced by Şimşek (2009) as a new approach to the Subjective Well-Being (SWB) perspective that exists in the fields of history, philosophy and psychology. The Ontological Well-Being Scale (OWBS), developed by Şimşek (2009) in accordance with this perspective, yielded significant results in positive and negative mental health areas, and was found to be related to the concepts of internal motivation and psychological well-being. The scale, which is grouped as "Past", "Now" and "Future", includes a total of 24 question items. The scale has four sub-dimensions: "nothingness" (meaninglessness), "activation" (activity), "regret" (regret) and "hope" (hope). The scale filled out based on my self-evaluation method was evaluated on a five-point scale; Participants are expected to mark an answer between "I don't feel at all" (1 point) and "I feel very intensely" (5 points) for each question.

SECONDARY OUTCOMES:
Beck Depression Scale | 8 Months
  The Beck Depression Scale was developed by Beck in 1961 to measure the risk of depression, the level of depressive symptoms and the change in severity in adults. The Turkish validity and reliability study was carried out by Hisli in 1989. Beck Depression Inventory is a 21-item self-assessment scale. Each item is related to a behavioral feature related to depression and is scored between 0 and 3 according to the severity of depression. The total score of the scale ranges from 0 to 63. If the score is between 0 and 9, there is no depression, 10-16 points indicate mild, 17-24 points indicate moderate, and 25 and higher points indicate severe depressive symptoms. Hisli (1989) calculated the reliability coefficient of the scale as 0.80 with the item analysis method and as 0.74 with the split-test method.

IPD SHARING:
Plan to Share IPD: No